CLINICAL TRIAL: NCT04238507
Title: A Clinical Study of the USASK Airway - An Improved Oral Airway for Bag-Mask Ventilation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, William McKay, Professor Emeritus, University of Saskatchewan
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Device Feasibility
Other Study IDs: BIO-1324
Record Dates: First submitted 2019-08-12; First posted 2020-01-23 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Anesthesia, General

STUDY DESIGN:
Intervention Model Description: : The proposed experiment is a repeated-measures unblinded randomized controlled trial (RCT), with randomization of the order of use, comparing BMV using a Guedel air or the UA device on the same participant.
Who Masked: Participant, Investigator
Masking Description: In the OR, the investigator will open an opaque numbered envelope with the randomization order for the performance of BMV.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guedel airway (OPA) (Active Comparator): Following induction of GA, air:O2 flows will be set at 0:10L, the Adjustable Pressure Limiting (APL) valve set to 50cm water pressure, and the reservoir bag filled. The learner will perform BMV with a Guedel airway placed by the anesthesiologist, while the anesthesiologist ensures that the reservoir bag is filled between breath attempts by using the oxygen flush.
  Interventions: Device: Guedel airway
- McKay Airway (MA) (Active Comparator): Following induction of GA, air:O2 flows will be set at 0:10L, the Adjustable Pressure Limiting (APL) valve set to 50cm water pressure, and the reservoir bag filled. The learner will perform BMV with a USASK airway placed by the anesthesiologist, while the anesthesiologist ensures that the reservoir bag is filled between breath attempts by using the oxygen flush.
  Interventions: Device: USASK airway

INTERVENTIONS:
Device: Guedel airway — Following induction of GA, air:O2 flows will be set at 0:10L, the Adjustable Pressure Limiting (APL) valve set to 50cm water pressure, and the reservoir bag filled. The learner will perform BMV with a Guedel airway placed by the anesthesiologist, while the anesthesiologist ensures that the reservoir bag is filled between breath attempts by using the oxygen flush.
  Arms: Guedel airway (OPA)
Device: USASK airway — Following induction of GA, air:O2 flows will be set at 0:10L, the Adjustable Pressure Limiting (APL) valve set to 50cm water pressure, and the reservoir bag filled. The learner will perform BMV with a USASK airway placed by the anesthesiologist, while the anesthesiologist ensures that the reservoir bag is filled between breath attempts by using the oxygen flush.
  Arms: McKay Airway (MA)

SUMMARY:
A clinical study of USASK AIRWAY - An Improved Oral Airway for Bag-mask Ventilation

A clinical study of MA AIRWAY - An Improved Oral Airway for Bag-mask Ventilation We report a study with University Research Ethics Board approval of a new oral airway device, the McKay Airway (MA), designed for easy maintenance of jaw-thrust (see illustration) for first responders who may perform bag-mask venti-lation (BMV) infrequently, and who often do not perform it well. Null hypothesis: naïve learners' time to achieve exhaled tidal volume (VE) >300ml will be no dif-ferent using MA than using a Guedel oropharyngeal airway (OPA) on anesthetized patients. Design was a repeated-measures unblinded controlled trial with blinded randomization of the order of airway use, comparing MA versus OPA conducted from July until December 2019. Anesthesiologists' decision to intervene and comments were recorded. Consenting learners included medical students, resi-dents from specialties other than anesthesiology, operating room staff, or naïve learners in technical courses scheduled in the operating rooms to be taught airway management. Patients were consenting adults booked for elective surgery under general anesthesia (GA). Excepted patients were those with loose incisors, tem-poromandibular joint disorders, reflux, those who did not wish to participate, and those whom the attending anesthesiologist felt put them at any added risk by par-ticipating. For patients with missing teeth, we padded the MA surface with 1cm thick stick-on sponge (Reston™ Self-Adhering Foam Pads; 3M, Maplewood MN USA). Patients were under the direct care of the consenting staff anesthesiologist for that OR. They were recruited in Pre-Admission Clinic, the hospital wards, Same-Day and Day-Surgery units, and in the OR holding area.

The experimental procedure included normal preoxygenation, induction of anesthesia, and BMV by the attending anesthesiologist as needed to assure high oxygen saturation prior to opening an opaque numbered envelope to randomly choose which airway to use first. We mimicked a self-inflating BMV device with the anesthetic machine by setting the Adjustable Pressure Limiting (APL) valve to >30cm water pressure and using the oxygen flush to ensure that the reservoir bag was filled between breath attempts. With the randomized airway in place, learners applied the mask with their left hand, squeezing the bag with their right approxi-mately every 3s. We timed from the first bag squeeze until VE exceeded 300ml, then repeated the experiment with the other airway. We approached 56 patients, recruited 34 female and 20 male, and obtained data for 51. One obese patient had severe succinylcholine fasciculations with rapid profound desaturation and the an-esthesiologist took over immediately, and for two the anesthesiologist misunder-stood the experiment. Time measurements were analysed with Wilcoxon's Signed Rank test, incidences with Fisher's Exact test or Chi Square. MA allowed faster adequate ventilation than OPA: Hodges-Lehmann median difference: 6s [95% CI 5 to 6.3s]; quartiles: OPA 9.5 to 37s; MA 7 to 16s range: OPA 5 to 78s; MA 2 to 49s; p = 0.02. When used first, the MA was faster than the OPA 30% of times compared to 11% when OPA was used first (p = 0.04), suggesting that MA may be easier to learn. Comments: 16 preferred the MA, 2 the OPA, and 15 had no preference (p = 0.02 compared to equal preferences). Further studies are warrant-ed.

DETAILED DESCRIPTION:
INTRODUCTION A newly invented airway device, the McKay Airway (MA) may improve ventilating a patient with a mask and self-inflating bag attached to an oxygen source (bag-mask ventilation: BMV), a common and often lifesaving step in anesthesia, intensive care, and emergency practice. BMV has been shown to frequently provide no or inadequate ventilation in the hands of beginners or those who practice it rarely; studies report successful BMV by beginners of 43 to 85%, with the latter requiring an average time of 44s to achieve successful ventilation. A study is proposed to assess the functionality of the device for BMV comparing MA with the widely used Guedel oropharyngeal airway (OPA). The MA does not cause gagging or vomiting in patients with a fluctuating level of consciousness.

Null hypothesis: Naïve learners will perform BMV no better using the new MA device than using a Guedel airway (current standard device in use for BMV) as measured by time to Vt > 300ml.

Design: Repeated-measures unblinded randomized controlled trial (RCT), with randomization of the order of use, comparing BMV using a Guedel air or the MA device on the same participant.

Primary outcome: Time from applying the mask to achieving ventilation with Vt > 300ml.

Secondary outcomes: An anesthesiologist's decision to intervene will be noted and counted should it occur. If there is adequate ventilation by 30s, the attempt will be considered a success; otherwise a failure. Scores will be recorded on rating scales for each BMV method: ease of insertion, ease of holding the mask properly, ease of obtaining a good seal, ease of obtaining an open airway, and likelihood of employing the method in practice. Comments about overall impression will be recorded.

Participants: Participants are of three kinds: learners, patients, and anesthesiologists. Learners will be consenting medical students, residents from specialties other than anesthesiology, or naïve learners in the Respiratory Technician or Emergency Medical Technician courses, all of whom are routinely rotated through the Saskatoon operating rooms (ORs) to learn airway management. Excepted will be learners who do not wish to participate. Patients will be consenting adult (age ≥ 18 years) patients booked into the operating rooms of SHR for elective surgery under general anesthesia (GA). BMV is normal clinical practice for all patients as part of the induction and emergence phases of GA. Excepted patients will be those with temporomandibular joint disorders, those who do not wish to participate, those whom the attending anesthesiologist feels puts them at any added risk by participating, and those whose anesthetic plan is changed from GA to a regional anesthetic technique. They will be under the direct constant care of the consenting staff anesthesiologist for that OR. Excepted anesthesiologists will be those who do not wish to participate in the study in general or for any particular patient or operation.

Number of participants: Sample size calculation for repeated measures t-test with effect size 0.33, alpha 0.05, power 0.8 is 59. We will recruit 65 to 80 for logistical OR exigencies.

Consent: With University of Saskatchewan Research Ethics Board approval, investigators, will recruit learners, anesthesiologists, and patients. Patients will be recruited in Pre-Admission Clinic (PAC), on the hospital wards, in Same-Day and Day-Surgery units, and in the OR holding area.

Data and privacy concerns will accord with University of Saskatchewan Ethics Committee principles.

Patient safety: The experiment will be overseen by the attending specialist anesthesiologist who will intervene immediately as needed and proceed as clinically indicated if even the smallest issue of patient safety arises during learners' attempts at BMV. This is not different from the normal clinical teaching situation. Risk to participating patients is minimal.

Interventions: Prior to their rotation in the ORs, consenting learners will watch teaching videos to learn BMV using OPA and MA.

Statistical analysis. Demographic data will be tabulated as observational. Time measurements will be tested for normality by Shapiro-Wilk, and if passed, by paired t-test; otherwise by Wilcoxon Signed Rank Test. Incidence data will be compared by Fishers Exact test or Chi-squared.

ELIGIBILITY:
Inclusion Criteria: Participants are of three kinds: learners, patients, and anesthesiologists. Learners will be consenting medical students, residents from specialties other than anesthesiology, or naïve learners in the Respiratory Technician or Emergency Medical Technician courses, all of whom are routinely rotated through the Saskatoon operating rooms (ORs) to learn airway management. Excepted will be learners who do not wish to participate. Patients will be consenting adult (age ≥ 18 years) patients booked into the operating rooms of SHR for elective surgery under general anesthesia (GA). BMV is normal clinical practice for all patients as part of the induction and emergence phases of GA -

Exclusion Criteria: Excepted patients will be those with temporomandibular joint disorders, those who do not wish to participate, those whom the attending anesthesiologist feels puts them at any added risk by participating, and those whose anesthetic plan is changed from GA to a regional anesthetic technique

-

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2019-07-22 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Time from applying the mask to achieving ventilation | 1 minute
  Time from applying the mask to achieving ventilation with tidal volume >300ml.

SECONDARY OUTCOMES:
airway use questions | 15 minutes
  An anesthesiologist's decision to intervene and take over BMV will be noted and counted should it occur. If there is adequate ventilation by 30s, the attempt will be considered a success; otherwise a failure. Scores will be recorded on rating scales for each BMV method: ease of insertion, ease of holding the mask properly, ease of obtaining a good seal, ease of obtaining an open airway, and likelihood of employing the method in practice. Comments about overall impression will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Gamble, Study Director — University of Saskatchewan Dept. of Anesthesia Research Director
Locations (1):
- Saskatoon Health Region, 410 22nd Street East, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No